CLINICAL TRIAL: NCT01480063
Title: A Multicenter, Multinational, Observational Study to Collect Information on Safety and to Document the Drug Utilization of Fampyra® When Used In Routine Medical Practice (LIBERATE)
Brief Title: An Observational Study to Collect Information on Safety and to Document the Drug Utilization of Fampyra (BIIB041) When Used In Routine Medical Practice
Acronym: LIBERATE
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 218MS401
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Fampyra: Fampyra administered as prescribed in routine clinical practice.
  Interventions: Drug: Fampridine

INTERVENTIONS:
Drug: Fampridine — Fampridine administered as prescribed in routine clinical practice. Biogen is not supplying drug for this study.
  Other Names: Ampyra; dalfampridine; Fampyra; BIIB041; fampridine prolonged-release tablets

SUMMARY:
The primary objective of the study is to collect additional safety data including the incidence rate of seizure and other specific Adverse Events (AEs) of interest from participants taking Fampyra in routine clinical practice. The secondary objectives of this study are to characterize utilization patterns of Fampyra in routine clinical practice, to assess the effectiveness of risk minimization measures as described in the risk management plan for Fampyra, to assess the change over time in participant self-reported evaluation of the physical and psychological impact of Multiple Sclerosis (MS) while taking Fampyra and to assess the change over time in physician assessment of walking ability in participants taking Fampyra (MS participants only).

ELIGIBILITY:
Key Inclusion Criteria:

* MS patients with any disease subtype who are ≥18 years of age and must have been newly prescribed Fampyra but not yet started the treatment.
* Patients who are willing and able to provide written informed consent.

Key Exclusion Criteria:

* None

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This post marketing study will be carried out by neurologists in routine clinical settings.
Sampling Method: Non-Probability Sample
Enrollment: 4734 (Actual)
Dates: Start 2012-04-16 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Day 1 up to one year

SECONDARY OUTCOMES:
Utilization patterns of Fampyra in Routine Clinical Practice | Day 1 up to one year
  Variables to be characterized include reason for Fampryra use, dose and duration of use, dosing deviations from local Fampyra label, and reasons for dosage changes.
Effectiveness of risk minimization measures | Day 1 up to one year
  Variables to be characterized may include demographics, medical history, reasons for Fampyra use, dose deviation from local Fampyra label and overdoses.
Change from Baseline in Physician's Clinical Global Impression of Improvement (CGI-I) of Walking Ability Assessed Whenever the Multiple Sclerosis Participant is Seen by the Neurologist | Baseline, Day 1 up to one year
  The Clinical Global Impression-Improvement (CGI-I) scale is a 7-point scale that requires the clinician to rate the improvement or worsening of the overall walking ability of the patient.
Participants' Assessment of Physical and Psychological Impact of Multiple Sclerosis Using the Multiple Sclerosis Impact Scale-29 Items (MSIS-29) | Baseline, Months 3, 6, 9, 12
  The 29-item Multiple Sclerosis Impact Scale (MSIS-29) is a patient-reported outcome measure to assess the impact of MS on day-to-day life during the past 2 weeks from a patient's perspective; it measures 20 physical items and 9 psychological items. The physical score is generated by summing individual items and then transforming to a scale with a range of 0 to 100, where high scores indicate worse health.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (164):
- Argentina (5):
  - Research Site, Ciudad Autonoma de Buanos Aires, Buenos Aires
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research Site, Salta
- Canada (6):
  - Research Site, Burnaby, British Colombia
  - Research Site, Fredericton, New Brunswick
  - Research Site, Brampton, Ontario
  - Reasearch Center, London, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
- Czechia (4):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Pardubice
  - Research Site, Prague
- France (42):
  - Research Site, Agen, Lot Et Garonne
  - Research Site, Rouen, Sein Maritime
  - Research Site, Bois-Guillaume, Seine-Maritime
  - Research Site, Angers
  - Research Site, Bayonne
  - Research Site, Bordeaux
  - Research Site, Bron
  - Research Site, Caen
  - Research Site, Cahors
  - Research Site, Cergy
  - Research Site, Colmar
  - Research Site, Dax
  - Research Site, Dijon
  - Research Site, Gonesse
  - Research Site, La Seyne-sur-Mer
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lisieux
  - Research Site, Lyon
  - Research Site, Mantes-la-Jolie
  - Research Site, Marseille
  - Research Site, Montauban
  - Research Site, Montbéliard
  - Research Site, Montluçon
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Pringy
  - Research Site, Quimper
  - Research Site, Rambouillet
  - Research Site, Roanne
  - Research Site, Rouen
  - Research Site, Rueil-Malmaison
  - Research Site, St-Malo
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Vichy
- Germany (48):
  - Research Site, Sindelfingen, Baden-Wurttemberg
  - Research Site, Karlstadt am Main, Bavaria
  - Research Site, Lohr a. Main, Bavaria
  - Research Site, Munich, Bavaria
  - Research Site, Neusäß, Bavaria
  - Research Site, Göttingen, Lower Saxony
  - Research Site, Wermsdorf, Nordsachsen
  - Research Site, Homburg, Saarland
  - Research Site, Stadtroda, Thuringia
  - Research Site, Abensberg
  - Research Site, Altenholz
  - Research Site, Aschaffenburg
  - Research Site, Bad Krozingen
  - Research Site, Bamberg
  - Research Site, Bayreuth
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bogen
  - Research Site, Bonn
  - Research Site, Butzbach
  - Research Site, Eisenach
  - Research Site, Erbach im Odenwald
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Grevenbroich
  - Research Site, Hagen
  - Research Site, Hamburg
  - Research Site, Herford
  - Research Site, Itzehoe
  - Research Site, Kastellaun
  - Research Site, Landshut
  - Research Site, Lappersdorf
  - Research Site, Leipzig
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Neu-Ulm
  - Research Site, Neuburg am Inn
  - Research Site, Oldenburg
  - Research Site, Ostfildern
  - Research Site, Ravensburg
  - Research Site, Singen
  - Research Site, Sinsheim
  - Research Site, Stade
  - Research Site, Stuttgart
  - Research Site, Trier
  - Research Site, Ulm
  - Research Site, Unterhaching
- Research Site, Dublin, Ireland
- Israel (3):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Tel Aviv
- Research Site, Beirut, Lebanon
- Netherlands (25):
  - Research Site, Almelo
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Blaricum
  - Research Site, Breda
  - Research Site, Dordrecht
  - Research Site, Eindhoven
  - Research Site, Emmen
  - Research Site, Enschede
  - Research Site, Flushing
  - Research Site, Gouda
  - Research Site, Groningen
  - Research Site, Heerenveen
  - Research Site, Hoorn
  - Research Site, Leeuwarden
  - Research Site, Leiden
  - Research Site, Meppel
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Sittard Geleen
  - Research Site, Sneek
  - Research Site, Tilburg
  - Research Site, Venlo
  - Rsearch Site, Zutphen
- Norway (3):
  - Research Site, Bergen
  - Research Site, Molde
  - Research Site, Stavanger
- Portugal (9):
  - Research Site, Amadora
  - Research Site, Braga
  - Research Site, Faro
  - Research Site, Guimarães
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Matosinhos Municipality
  - Research Site, Porto
  - Research Site, Viana do Castelo
- Spain (15):
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Getafe, Madrid
  - Research Site, Pamplona, Navarre
  - Research site, San Cristóbal de La Laguna, Tenerife
  - Site Research, Bilbao, Vizcaya
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Ávila
  - Research Site, Cáceres
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Segovia
  - Research Site, Valladolid
  - Research Site, Zaragoza
- United Arab Emirates (2):
  - Research Site, Abu Dhabi
  - Research Site, Dubai

REFERENCES:
- [Derived] Castelnovo G, Gerlach O, Freedman MS, Bergmann A, Sinay V, Castillo-Trivino T, Kong G, Koster T, Williams H, Gafson AR, Killestein J. Safety, Patient-Reported Well-Being, and Physician-Reported Assessment of Walking Ability in Patients with Multiple Sclerosis for Prolonged-Release Fampridine Treatment in Routine Clinical Practice: Results of the LIBERATE Study. CNS Drugs. 2021 Sep;35(9):1009-1022. doi: 10.1007/s40263-021-00840-x. Epub 2021 Jul 28. PMID 34322853